CLINICAL TRIAL: NCT07060690
Title: A Women-Centered Approach: Evaluating a Human-Supported Online Intervention for Depression. Study on Its Efficacy and the Metabolic Signature of Personalised Treatment Response
Brief Title: Evaluating a Personalised Online Program With Human Support for Women With Depression and Its Impact on Mental Health and Biological Changes
Acronym: 3D01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Francesc Colom, PsyD, PhD (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Hospital del Mar (Other)
Responsible Party: Sponsor-Investigator, Francesc Colom, PsyD, PhD, Principal Investigator, Hospital del Mar Research Institute (IMIM)
Organization: Hospital del Mar Research Institute (IMIM) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PI23/00257; 2023/11236/I (Other: Hospital del Mar Drug Research Ethical Committee (CEIm))
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Depression Symptoms; Depression - Major Depressive Disorder; Depressive Disorder
Keywords: Women; Metabolomics; Depression; Internet-Based Intervention; Personalized Medicine
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Other key personnel, including clinicians, statisticians, lab technicians in the Metabolomics Unit, and the principal investigator, will remain blind to the randomisation procedure and group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Internet-based Cognitive Behavioural Therapy (iCBT) with human interaction+ Treatment as usual (TAU) (Experimental): Participants will undertake the 3D programme, a 10-week internet-delivered cognitive behavioural therapy (iCBT) intervention tailored for women.
  Interventions: Behavioral: iCBT with human interaction
- Brief psychoeducational videos + TAU (Active Comparator): Participants will continue to receive their usual treatment for depression from their healthcare team throughout the study. Additionally, over 10 weeks, they will receive biweekly emails containing links to six brief educational video capsules covering depression causes, behavioural activation, hormonal cycle effects, sleep strategies, healthy habits, and relapse prevention.
  Interventions: Behavioral: Psychoeducational videos

INTERVENTIONS:
Behavioral: iCBT with human interaction — The 3D programme is a 10-week online intervention based on Cognitive Behavioural Therapy (CBT), designed to support women's mental health. Participants will use the 3D website to complete 10 weekly self-guided modules that include videos, written materials, and interactive activities. Topics address depression and issues commonly experienced by women, such as hormonal changes, caregiving, body image, and sexism. All content is available in both video and text formats. Participants will also have six one-to-one video sessions with a trained health/clinical psychologist, who will tailor the programme by recommending specific modules or tasks. All therapists will complete training on the 3D programme and online therapy. Participants will receive guidance on how to use the 3D website before starting.
  Other Names: 3D
  Arms: Internet-based Cognitive Behavioural Therapy (iCBT) with human interaction+ Treatment as usual (TAU)
Behavioral: Psychoeducational videos — This control arm provides psychoeducational content without therapist support or homework assignments, serving as an adjunct to standard care. This distinguishes it from the experimental arm, which includes therapist-guided interventions and active homework components.
  Arms: Brief psychoeducational videos + TAU

SUMMARY:
This study aims to evaluate the efficacy of a specially developed internet-based Cognitive Behavioural Therapy (CBT) programme with human interaction-referred to as the 3D programme-tailored specifically for women experiencing mild to moderate depressive symptoms. We hypothesise that participation in the intervention will lead to greater improvements in depression severity, compared to receiving only brief psychoeducational videos, when used as an add-on to treatment as usual (TAU) in this population.

The 3D programme is a 10-week blended intervention that includes ten weekly online self-guided modules focused on depression and women's health, along with six individual video sessions with a health/clinical psychologist. The modules cover topics such as mood changes across the menstrual cycle, body image, stress, caregiving, and the impact of gender-based experiences on mental health.

To explore how biological factors may influence how participants respond to treatment, the study will collect biological samples. These will be analysed to track hormone and metabolic changes, with the goal of identifying biological markers that might predict who benefits most from the intervention.

Ultimately, the results of this study aim to improve access to effective and personalised mental health care for women by evaluating whether a structured and personalised online CBT programme can provide meaningful benefits.

DETAILED DESCRIPTION:
OBJECTIVES Primary objective: To assess the impact of the 3D programme on depressive symptom severity compared to a psychoeducational control condition.

Secondary objectives: To evaluate improvements in overall functioning, quality of life, perceived stress, and menstruation-related distress. Additionally, the study will investigate metabolic signatures associated with treatment response, focusing on tryptophan and steroid hormone pathways.

HYPOTESES Main hypothesis: Participation in the 3D programme will lead to greater improvements in depression severity (measured by HDRS-17) compared to receiving only informational materials when used as an add-on to Treatment As Usual (TAU) in women experiencing mild to moderate depressive episodes.

Secondary hypotheses:

1. Participation in the 3D programme will improve overall functioning in women with mild to moderate depressive episodes.
2. Participation in the 3D programme will improve health-related quality of life in women with mild to moderate depressive episodes.
3. Participants in the 3D programme with higher perceived stress levels will show less improvement in depression severity compared to those with lower stress levels.
4. Participants in the 3D programme with higher menstruation-related distress will show greater improvement in depression severity than those with lower levels of distress.
5. Participants in the 3D programme with more gynaecological problems will experience greater improvement in depression severity than those with fewer gynaecological issues.
6. A metabolic signature related to tryptophan metabolism and steroid hormones will predict the response to the 3D intervention.
7. Participation in the 3D programme will lead to changes in hormone production and/or balance, with the persistence of these hormonal changes correlating with the long-term effects of the intervention.

SAMPLE SIZE ESTIMATION AND RECRUITMENT The optimal sample size is estimated to be 60 participants per group. This calculation is based on a Cohen's d effect size of 0.2, a 95% confidence interval, a statistical power of 90%, and an anticipated attrition rate of 20%. Sample size estimation was conducted using G* Power 3.1.7 software.

All patients meeting the inclusion and exclusion criteria will be invited to participate in the study by their treating team at the outpatient mental health facilities within Hospital del Mar. Additionally, gynaecologists at Hospital del Mar will be encouraged to refer patients suspected of experiencing depressive symptoms. In such cases, patients will be screened by the study psychologist/psychiatrist to confirm these symptoms. Recruitment will conclude upon reaching the target of 120 participants with complete data.

RANDOMISATION AND BLINDING Participants will be randomised in a 1:1 ratio using the REDCap randomisation module, which will automatically assign participants to either the experimental or control group through simple randomisation with equal allocation.

This study will implement single blinding. Due to the nature of the intervention, participants will be aware of their group assignment (experimental or control) following randomisation. Likewise, therapists delivering the intervention will be aware of the assigned group, as is standard practice in psychological intervention trials. To uphold the integrity of the blinding process, the following measures will be applied:

1. Personnel responsible for data analysis will remain blinded to group assignments.
2. Independent raters conducting outcome assessments will be blinded to participant group allocation.
3. Other stakeholders, including clinicians, statisticians, and the principal investigator, will remain unaware of the randomisation process and group assignments to minimise potential bias.

STUDY DESING Part 1. Randomised controlled trial The study follows a naturalistic treatment approach, ensuring that all participants continue their usual care. The study will be conducted in accordance with the CONSORT guidelines.

PART 2. Metabolic signature of treatment response The metabolic signature of treatment response will be characterised through the analysis of tryptophan and steroid-related pathways. All analyses will be conducted using methods developed and validated by the Applied Metabolomic Research Group at Hospital del Mar Research Institute, ensuring proper sample handling protocols as outlined in previous studies.

Tryptophan Metabolism:

Tryptophan pathway metabolites-including tryptophan, kynurenine, serotonin, 3-hydroxykynurenine, 5-hydroxyindoleacetic acid, and kynurenic acid-will be quantified using liquid chromatography-tandem mass spectrometry (LC-MS/MS). The analysis will follow the protocol established by Marcos et al.

Analysis will focus on the kynurenine/tryptophan (K/T) ratio, a marker of indoleamine-2,3-dioxygenase (IDO) activity, which plays a key role in immune regulation and inflammatory responses.

Additionally, serotonin synthesis and its relationship with tryptophan availability will be assessed, alongside the tryptophan/large neutral amino acid (LNAA) ratio, which serves as an indicator of tryptophan's availability for serotonin production. Data will be integrated using network analysis to identify potential associations between these metabolites and treatment response.

Steroid Hormones:

The steroid profile will be analysed to monitor key sex hormones (e.g., estradiol, testosterone, progesterone) and glucocorticoids (e.g., cortisol, 20α-DHE, and 20β-DHE), along with their metabolites. These hormones play a pivotal role in modulating inflammation and metabolic pathways, with altered levels linked to physiological stress responses and treatment outcomes. These measurements will be performed by LC-MS/MS, following the method previously outlined by the research group.

Biological Samples:

Analysis will be conducted using various biological matrices, including blood, saliva, urine, nails, and hair, to provide complementary insights. Saliva, blood, and urine samples will capture acute metabolic changes at the time of the visit, while nails and hair will reflect chronic metabolite production.

ASSESSMENTS Assessments will be carried out at baseline (T0), immediately following the intervention (3 months after baseline, T1), and at a follow-up assessment (6 months after baseline, T2).

The baseline assessment will include:

* Collection of socio-demographic and clinical data, with self-reported information gathered via a secure, online-based assessment system (REDCap).
* Collection of biological samples (blood, saliva, urine, nails, and hair), with sample collection times recorded to account for circadian-sensitive metabolites. These samples will be collected exclusively from cisgender women.
* A gynaecology consultation to assess hormonal and menstrual complications. These will be evaluated using a 5-point Likert scale, ranging from "1 - No complication" to "5 - Severe complication requiring significant gynaecological intervention or further medical examination." Patients who require additional medical evaluations will be referred for appropriate follow-up care.
* Metabolic analysis, focusing on tryptophan metabolism and steroid hormone regulation, with the goal of identifying biomarkers predictive of therapeutic outcomes.

Clinical data and biological samples will be collected at all time points.

DATA MANAGEMENT All the data will be text-based (.docx) or numeric format (.xlsx). For all published files, a document record and change track will be included (author contact information, status, version, change reason and date, contents" description, title, origin of the data including a description of the measurement and/or experiment setup) in a separate metadata file for each characterization action called METADATA.ODS.

Data will be stored on a secure server at the Hospital del Mar Research Institute, in compliance with EU and Spanish data protection regulations (General Data Protection Regulation, GDPR, of May 25, 2018; and Organic Law 3/2018 of December 5, on the Protection of Personal Data and Guarantee of Digital Rights).

STATISTICAL ANALYSIS

Primary and Secondary Outcomes:

Analyses will follow an intention-to-treat (ITT) approach, including all participants according to their randomized allocation, regardless of adherence to the intervention.group. Linear mixed-effects models (LMMs) will be used to examine changes over time and between groups for the HDRS-17, WHO-DAS 2.0, EQ-5D-5L, PSS, and MEDI-Q scores. These models will include fixed effects for group, time, and their interaction, and a random intercept for participants to account for within-subject correlation over time. Where appropriate, subscale-level analyses and models using change scores will also be conducted for secondary outcomes. To further explore the temporal dynamics of the intervention's effects, post hoc simple effects analyses will be performed to probe significant interactions.

Additional Analyses:

LLMs and multiple linear regression models will be employed to identify predictors of clinical improvement. Additionally, moderator analyses using linear mixed models will assess whether levels of perceived stress (PSS), or menstrual distress (MEDI-Q) influence treatment response as measured by changes in HDRS-17 scores over time.

Exploratory Biomarker Analyses:

Partial Least Squares Regression (PLSR) and multiple regression will be conducted to model associations between metabolite profiles, their changes over time, and changes in depressive symptoms. Variable Importance in Projection (VIP) scores and cross-validation techniques will be applied to evaluate model performance and identify key predictive biomarkers. Additionally, metabolomic evolution will be assessed through exploratory factor analysis, grouping variables into latent factors.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Age between 18 and 45 years (inclusive)
* Mild to moderate depressive symptoms, defined by a score of 17 to 23 on the 17-item Hamilton Depression Rating Scale (HDRS-17)
* Fluent in Spanish
* Access to the internet and the ability to use digital devices (e.g., smartphone, tablet, or computer)

Exclusion Criteria:

* Currently receiving psychological therapy
* Participation in any other interventional clinical trial for depression within the past 3 months
* Pregnant or planning to become pregnant during the study period
* Cognitive impairment that may interfere with informed consent or study participation
* Presence of psychotic symptoms, active suicidal ideation, or current substance abuse disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Depression severity | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline
  Change in depressive symptoms, as measured by the 17-item Hamilton Depression Rating Scale (HDRS-17), validated in Spanish. Score range: 0 to 52; higher scores indicate more severe depression.

SECONDARY OUTCOMES:
Overall functioning | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline
  Change in overall functioning, measured using the World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS 2.0, 36-item version), self-administered and validated in Spanish.The WHO-DAS 2.0 assesses functioning across six domains. Higher scores indicate greater disability. The Spanish version has demonstrated strong psychometric properties across psychiatric populations.
Health-related quality of life | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline.
  Change in health-related quality of life, assessed using the EQ-5D-5L, a self-reported questionnaire validated in Spanish.
  The EQ-5D-5L measures five dimensions. Each dimension is rated on a 5-point scale, and responses are combined into a single index score ranging from below 0 (very poor health) to 1 (perfect health). Additionally, a Visual Analogue Scale (VAS) is included, ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Perceived Stress | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline.
  Change in perceived stress, measured using the Perceived Stress Scale (PSS-10), a 10-item self-reported questionnaire validated in Spanish.
  Each item is rated on a 5-point scale from 0 (never) to 4 (very often). Total scores range from 0 to 40, with higher scores indicating greater levels of perceived stress.
Menstruation-related distress | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline.
  Change in menstruation-related distress, measured using the Menstrual Distress Questionnaire (MEDI-Q), a 25-item self-reported tool assessing symptoms such as pain, discomfort, psychological changes, gastrointestinal issues, and physiological alterations.
  The MEDI-Q is a novel instrument and does not yet have a validated Spanish version; this study may contribute to its adaptation for Spanish-speaking populations.

OTHER OUTCOMES:
Tryptophan metabolism biomarkers | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline.
  Quantification of tryptophan and related metabolites (kynurenine, serotonin, 3-hydroxykynurenine, 5-hydroxyindoleacetic acid, kynurenic acid) and calculation of metabolic ratios (e.g., kynurenine/tryptophan ratio) using LC-MS/MS in biological samples (blood, saliva, urine, nails, hair). Higher or altered levels may be associated with treatment response.
Steroid hormone profile | Baseline (T0): At enrolment/start of intervention. Post-intervention (T1): 3 months after baseline. Follow-up (T2): 6 months after baseline.
  Changes in hormone production and balance over time associated with intervention participation. Measurement of sex hormones (estradiol, testosterone, progesterone) and glucocorticoids (cortisol, 20α-DHE, 20β-DHE) and their metabolites using LC-MS/MS in biological samples (blood, saliva, urine, nails, hair). Hormonal alterations over time will be evaluated as potential markers of treatment effects.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar Research Institute, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Vannuccini S, Rossi E, Cassioli E, Cirone D, Castellini G, Ricca V, Petraglia F. Menstrual Distress Questionnaire (MEDI-Q): a new tool to assess menstruation-related distress. Reprod Biomed Online. 2021 Dec;43(6):1107-1116. doi: 10.1016/j.rbmo.2021.08.029. Epub 2021 Oct 26. PMID 34753680
- [Background] Remor E. Psychometric properties of a European Spanish version of the Perceived Stress Scale (PSS). Span J Psychol. 2006 May;9(1):86-93. doi: 10.1017/s1138741600006004. PMID 16673626
- [Background] Vazquez-Barquero JL, Vazquez Bourgon E, Herrera Castanedo S, Saiz J, Uriarte M, Morales F, Gaite L, Herran A, Ustun TB. [Spanish version of the new World Health Organization Disability Assessment Schedule II (WHO-DAS-II): initial phase of development and pilot study. Cantabria disability work group]. Actas Esp Psiquiatr. 2000 Mar-Apr;28(2):77-87. Spanish. PMID 10937388
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Ramos-Brieva JA, Cordero-Villafafila A. A new validation of the Hamilton Rating Scale for Depression. J Psychiatr Res. 1988;22(1):21-8. doi: 10.1016/0022-3956(88)90024-6. PMID 3397906
- [Background] Zimmerman M, Martinez JH, Young D, Chelminski I, Dalrymple K. Severity classification on the Hamilton Depression Rating Scale. J Affect Disord. 2013 Sep 5;150(2):384-8. doi: 10.1016/j.jad.2013.04.028. Epub 2013 Jun 4. PMID 23759278
- [Background] Krieger T, Bur OT, Weber L, Wolf M, Berger T, Watzke B, Munder T. Human contact in internet-based interventions for depression: A pre-registered replication and meta-analysis of randomized trials. Internet Interv. 2023 Mar 31;32:100617. doi: 10.1016/j.invent.2023.100617. eCollection 2023 Apr. PMID 37273939
- [Background] Marx W, McGuinness AJ, Rocks T, Ruusunen A, Cleminson J, Walker AJ, Gomes-da-Costa S, Lane M, Sanches M, Diaz AP, Tseng PT, Lin PY, Berk M, Clarke G, O'Neil A, Jacka F, Stubbs B, Carvalho AF, Quevedo J, Soares JC, Fernandes BS. The kynurenine pathway in major depressive disorder, bipolar disorder, and schizophrenia: a meta-analysis of 101 studies. Mol Psychiatry. 2021 Aug;26(8):4158-4178. doi: 10.1038/s41380-020-00951-9. Epub 2020 Nov 23. PMID 33230205
- [Background] Montcusi B, Madrid-Gambin F, Pozo OJ, Marco S, Marin S, Mayol X, Pascual M, Alonso S, Salvans S, Jimenez-Toscano M, Cascante M, Pera M. Circulating metabolic markers after surgery identify patients at risk for severe postoperative complications: a prospective cohort study in colorectal cancer. Int J Surg. 2024 Mar 1;110(3):1493-1501. doi: 10.1097/JS9.0000000000000965. PMID 38116682
- [Background] Marcos J, Renau N, Valverde O, Aznar-Lain G, Gracia-Rubio I, Gonzalez-Sepulveda M, Perez-Jurado LA, Ventura R, Segura J, Pozo OJ. Targeting tryptophan and tyrosine metabolism by liquid chromatography tandem mass spectrometry. J Chromatogr A. 2016 Feb 19;1434:91-101. doi: 10.1016/j.chroma.2016.01.023. Epub 2016 Jan 14. PMID 26818237
- [Background] Marcos J, Renau N, Casals G, Segura J, Ventura R, Pozo OJ. Investigation of endogenous corticosteroids profiles in human urine based on liquid chromatography tandem mass spectrometry. Anal Chim Acta. 2014 Feb 17;812:92-104. doi: 10.1016/j.aca.2013.12.030. Epub 2014 Jan 3. PMID 24491769